CLINICAL TRIAL: NCT03180411
Title: Colorectal Cancer Surveillance Decision Support Tool: Cognitive and Pilot Testing
Brief Title: Colorectal Cancer (CRC) Surveillance Tool: Cognitive and Pilot Testing
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PA16-0825; CE-1304-6855 (Other Grant/Funding Number: PCORI); NCI-2021-09747 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2017-06-02; First posted 2017-06-08 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; CRC; Colorectal cancer surveillance; Decision support tool; Interviews; Questionnaire; Survey
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cognitive Testing Phase Group: Participants take part in one-on-one interview with research staff and asked questions about participant's health and the disease.
  Interventions: Behavioral: Interview
- Pilot Testing Phase Group: After Cognitive Testing Phase interview, participants may be asked to have a second one-on-one interview with research staff.
  Participants may also be asked to complete a questionnaire about the disease, what participant understands about it, and the treatment plan recommended. Participant also asked to give participant's opinion about colorectal cancer follow-up materials.
  Interventions: Behavioral: Interview; Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Interview — Cognitive Testing Phase Group: Participants take part in one-on-one interview with research staff and asked questions about participant's health and the disease. The interview may take from 45-60 minutes to complete.
  Pilot Testing Phase Group: After Cognitive Testing Phase interview, participants have a second one-on-one interview. The interview will last from 45-60 minutes.
Behavioral: Questionnaire — Participant completes a questionnaire about the disease, what participant understands about it, and the treatment plan recommended. Participant asked to give participant's opinion about colorectal cancer follow-up materials. The questionnaire will take 35-45 minutes.
  Other Names: Survey
  Groups: Pilot Testing Phase Group

SUMMARY:
The goal of this research study to help develop a tool to assist patients in making decisions about care during treatment for colorectal cancer. Information collected during this study will be saved to help develop future studies about patient decision making in cancer treatment.

DETAILED DESCRIPTION:
Cognitive Testing Phase:

If participant agrees to take part in this study, participant will take part in a one-on-one interview where participant will be asked questions about participant's health and the disease. This is called the cognitive testing phase. Notes about the interviews may be kept so that the responses can be reviewed later by the study doctor and research staff.The interview may take from 45-60 minutes to complete.

Pilot Testing Phase:

Participant may be asked to take part in the next phase of the study called the pilot testing phase. If participant takes part in this phase, participant will have a second one-on-one interview. The interview will last from 45-60 minutes.

Participant may also be asked to complete a questionnaire about the disease, what participant understands about it, and the treatment plan recommended for participant. Participant will also be asked to give participant's opinion about colorectal cancer follow-up materials. If participant is asked to complete it, the questionnaire will be completed during the interview, in person. The questionnaire will take 35-45 minutes.

Collection of Information:

Information may be collected from participant's medical record about participant's health, participant's treatment, basic information like participant's age and participant's gender, and the disease. Information will not be collected from all participants.

Length of Study Participation:

If participant takes part in the cognitive testing phase only, participation in this study will end when participant has completed the interview.

If participant takes part in the pilot testing phase, participation in this study will end when participant has completed the second interview and questionnaire if participant was asked to complete it.

This is an investigational study.

Up to 100 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Able to read and speak English
3. Patient undergoing follow-up for curative resection of stage I-IV colon or rectal cancer
4. There will be no exclusion on the basis of gender or race.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal surgery clinics at UT MD Anderson Cancer Center in Houston, Texas
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Development of Decision Tool to Guide Participants in Making Individualized Decisions Regarding Colorectal Cancer (CRC) Surveillance Through the Use of Cognitive Testing Interviews | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: George Chang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org